CLINICAL TRIAL: NCT02663089
Title: An Open-label Study in Healthy Male Subjects, to Determine the Excretion Balance and Pharmacokinetics of [14C]-GSK961081, Administered as a Single Intravenous Microtracer (Concomitant With an Inhaled Non-radiolabelled Dose) and a Single Oral Dose
Brief Title: A Phase 1 (Ph1), Single Dose (SD), GSK961081 Absorption, Distribution, Metabolism, and Excretion (ADME) Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: Hammersmith Medicines Research (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201003
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: total radioactivity; [14C]-GSK961081; Pharmacokinetics; Chronic Obstructive Pulmonary Disease (COPD); Microtracer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Infusions, Intravenous; Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-GSK961081 IV+GSK961081 inhalation; [14C]-GSK961081 oral (Experimental): On Day 1 of Treatment Period 1, after an overnight fast of at least 8 hours, each subject will receive [14C] GSK961081 4 micrograms (mcg) by IV infusion over 1 hour. Within 5 minutes after the start of infusion, subjects will take 1200 mcg non-radiolabelled GSK961081 by inhalation. After Treatment Period 1, there will be a washout of at least 2 weeks. On Day 1 of Treatment Period 2, after an overnight fast of at least 8 hours, each subject will take 200 mcg [14C]-GSK961081 as an oral solution.
  Interventions: Drug: [14C]-GSK961081 solution for IV infusion; Drug: [14C]-GSK961081 oral solution; Drug: GSK961081 dry powder for inhalation

INTERVENTIONS:
Drug: [14C]-GSK961081 solution for IV infusion — Subjects will receive 10 mL of solution equivalent to 4 mcg of [14C]-GSK961081 (approximately 6.2 kilobecquerel [kBq]) intravenously as a single dose over 1 hour.
Drug: [14C]-GSK961081 oral solution — Subjects will receive 10 mL of solution equivalent to 200 mcg of [14C]-GSK961081 (approximately 311 kBq) orally as a single dose with up to 250 mL of water.
Drug: GSK961081 dry powder for inhalation — Subjects will receive single dose of 4 actuations of 300 mcg GSK961081 per actuation (1200 mcg GSK961081 total) as inhalation immediately after the start of infusion.

SUMMARY:
Batefenterol (GSK961081) is a bifunctional bronchodilator that is being developed for the treatment of Chronic Obstructive Pulmonary Disease (COPD). Absorption, metabolism and excretion of batefenterol have been studied in animals, in vitro, and in previous clinical studies; however, the elimination routes and metabolic pathways of batefenterol have not been fully elucidated in humans. This is an open-label, single centre, non-randomised, 2-period single-sequence crossover, mass balance study to determine total radioactivity (drug related material) in plasma, the rate and extent of excretion of total radioactivity in urine and faeces and the total recovery of radioactivity of [14C] GSK961081 administered as a single IV dose (concomitant with an inhaled non-radiolabelled dose) and a single oral dose, in healthy male subjects. A total of 6 healthy male subjects will be enrolled. The duration of each subject in the study is up to 11 weeks, which consists of a screening visit, 2 Treatment Periods, and a follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 30 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* A history of regular bowel movements (averaging one or more bowel movements per day).
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 19.0-31.0 kg/square metre (m^2) (inclusive)
* Sex: Male
* Subjects with female partners of child bearing potential must use a condom from the time of first dose of study medication until follow-up.
* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Mean corrected QT interval (QTc) > 450 milliseconds (msec)
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or 12-lead ECG.
* A pre-existing condition(s) interfering with normal gastrointestinal (GI) anatomy or motility, including constipation, malabsorption or other GI dysfunction which may interfere with the absorption, distribution, metabolism or elimination of the study drug. Subjects with a history of cholecystectomy must be excluded.
* At screening, a supine blood pressure (BP) that is persistently higher (triplicate measurements at least 2 min apart) than 140/90 millimetres of mercury (mmHg).
* At screening, a supine mean HR outside the range 40-90 beats per minute (BPM).
* Subject is mentally or legally incapacitated.
* A history of respiratory disease (e.g. history of asthmatic symptoms) in the last 10 years.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study medication, unless in the opinion of the investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >21 units. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 millilitres [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking; current smoker; or ex-smokers who gave up less than 6 months ago or who have a history of more than 10 pack-years. Pack-years = cigarettes per day multiplied by number of years smoked then divided by 20.
* History of sensitivity to any of the study medications or its components, or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates the subject's participation.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months before the first dose of study treatment.
* A positive test for Human Immunodeficiency Virus (HIV) antibody
* A positive pre-study drug/alcohol screen.
* The subject has participated in a clinical trial and has received an investigational product (IP) within 3 months before their first dose in the current study.
* Exposure to more than four new chemical entities within 12 months before the subject's first dose.
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months. A subjects' previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination/carryover into the current study.
* Subjects who have received a total body radiation dose of greater than 5.0 millisievert (mSv) (upper limit of World Health Organization [WHO] category II) or exposure to significant radiation (e.g. serial x ray or computed tomography [CT] scans, barium meal etc) in the 12 months before this study.
* An occupation which requires monitoring for radiation exposure, nuclear medicine procedures or excessive x-rays within the past 12 months.
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days before the first dose of study medication until the follow-up visit.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol, including the use of the enterotest capsule.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

PRIMARY OUTCOMES:
AUC(0 inf) of total drug-related material (radioactivity) in plasma after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25 , 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
  The following PK parameter will be measured: Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0 inf])
AUC(0-t) of total drug-related material (radioactivity) in plasma after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
  The following PK parameter will be measured: Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC[0-t]).
Cmax of total drug-related material (radioactivity) in plasma after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
  The following PK parameter will be measured: maximum observed plasma concentration (Cmax)
Tmax of total drug-related material (radioactivity) in plasma after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
  The following PK parameter will be measured: time of occurrence of Cmax (Tmax)
T1/2 of total drug-related material (radioactivity) in plasma after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
  The following PK parameter will be measured: terminal phase half-life (t1/2)
Volume of total radioactivity (drug related material) after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Clearance of total radioactivity (drug related material) after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Urinary and faecal cumulative excretion as a percentage of the total radioactive dose administered over time after a single IV microtracer of [14C] GSK961081 (concomitant with an inhaled non-radiolabelled dose) and a single oral dose of [14C] GSK961081 | Pre-dose and at 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-168 hours post-dose during Treatment Period 1 and 2

SECONDARY OUTCOMES:
AUC(0-inf) of parent GSK961081 and [14C] GSK961081 in plasma after a single IV microtracer of [14C]-GSK961081 concomitant with an inhaled non-radiolabelled GSK961081 dose and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
AUC(0-t) of parent GSK961081 and [14C] GSK961081 in plasma after a single IV microtracer of [14C]-GSK961081 concomitant with an inhaled non-radiolabelled GSK961081 dose and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Cmax of parent GSK961081 and [14C] GSK961081 in plasma after a single IV microtracer of [14C]-GSK961081 concomitant with an inhaled non-radiolabelled GSK961081 dose and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Tmax of parent GSK961081 and [14C] GSK961081 in plasma after a single IV microtracer of [14C]-GSK961081 concomitant with an inhaled non-radiolabelled GSK961081 dose and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
T1/2 of parent GSK961081 and [14C] GSK961081 in plasma after a single IV microtracer of [14C]-GSK961081 concomitant with an inhaled non-radiolabelled GSK961081 dose and a single oral dose of [14C] GSK961081 | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Volume of parent GSK961081 and [14C] GSK961081 after a single IV microtracer of [14C]-GSK961081 concomitant with an inhaled non-radiolabelled GSK961081 dose | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Clearance of parent GSK961081 and [14C] GSK961081 after a single IV microtracer of [14C]-GSK961081 concomitant with an inhaled non-radiolabelled GSK961081 dose | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Oral and inhaled absolute bioavailability (F) | Pre-dose and at 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96 and 168 hours post-dose during Treatment Period 1 and 2
Number of subjects with any adverse events (AEs) as a measure of safety | Up to 7 weeks
  An AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Composite of Hematology parameters as a measure of safety | Up to 11 weeks
  The following hematology parameters will be measured: Platelet Count, red blood cell (RBC) count, Hemoglobin, Hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), white blood cell (WBC) count, Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils
Composite of Clinical Chemistry parameters as a measure of safety | Up to 11 weeks
  The following clinical chemistry parameters will be measured: Urea, Creatinine, Glucose (fasting), Uric acid, Potassium, Sodium, Calcium, Chloride, phosphate, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Alkaline phosphatase, Gamma-glutamyl transferase (GGT), Cholesterol, Triglycerides, Total Bilirubin, Total Protein, Albumin, and Globulin.
Composite of Urinalysis parameters as a measure of safety | Up to 11 weeks
  The following urinalysis parameters will be measured by dip stick method: Protein, Blood, Ketones, glucose, bilirubin, urobilinogen, leukocyte esterase, specific gravity, nitrites, power of hydrogen (pH). If urine dipstick is abnormal for leukocyte esterase, nitrites, blood or protein, microscopic examination will be performed.
Electrocardiogram (ECG) as a measure of safety | Up to 11 weeks
  12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT using Bazett's formula (QTcB) or corrected QT using Fridericia's formula (QTcF) intervals.
Temperature as a measure of safety | Up to 11 weeks
Systolic and diastolic blood pressure as a measure of safety | Up to 11 weeks
Pulse rate as a measure of safety | Up to 11 weeks
Respiratory rate as a measure of safety | Up to 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Ambery C, Young G, Fuller T, Lazaar AL, Pereira A, Hughes A, Ramsay D, van den Berg F, Daley-Yates P. Pharmacokinetics, Excretion, and Mass Balance of [14 C]-Batefenterol Following a Single Microtracer Intravenous Dose (Concomitant to an Inhaled Dose) or Oral Dose of Batefenterol in Healthy Men. Clin Pharmacol Drug Dev. 2018 Nov;7(8):901-910. doi: 10.1002/cpdd.616. Epub 2018 Sep 19. PMID 30230263
- See also: Results for study 201003 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/201003?search=study&b'study_ids=201003'#rs